CLINICAL TRIAL: NCT01659957
Title: Behavioral Couples Group Therapy for Alcholic Patients: Clinical and Cost Outcomes
Brief Title: Couples Therapy for Alcoholic Patients
Acronym: CALM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Harvard University (Other)
Responsible Party: Principal Investigator, Timothy J. O'Farrell, Professor of Psychology, Harvard University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA017865 (NIH)
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Alcoholism
Keywords: Alcoholism; Couples
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group Couples Couseling (Experimental): Patients randomized to this arm will receive group couples counseling plus 12-step oriented alcoholism counseling.
  Interventions: Behavioral: Group Couples Counseling
- One-on-One Couples Couseling (Experimental): Patients randomized to this arm will receive one-on-one couples counseling plus 12-step oriented alcoholism counseling.
  Interventions: Behavioral: One-on-One Couples Counseling

INTERVENTIONS:
Behavioral: Group Couples Counseling
  Arms: Group Couples Couseling
Behavioral: One-on-One Couples Counseling
  Arms: One-on-One Couples Couseling

SUMMARY:
In treating alcoholism, many studies show Behavioral Couples Therapy (BCT) is more effective than typical counseling, but BCT is not widely used because standard BCT delivered one couple at a time is costly to deliver and does not fit with the primary group therapy focus of most community clinics. The proposed study will test with married or cohabiting alcoholic patients whether a group format for BCT will produce similar positive outcomes as standard BCT, and deliver these results at a lower cost. If outcomes are favorable, this could prompt clinics to start using group BCT and improve outcomes for alcoholic patients and their families.

DETAILED DESCRIPTION:
Multiple studies indicate that participation in Behavioral Couples Therapy (BCT) is associated with robust positive outcomes for alcoholic and drug-abusing patients, in terms of reduced substance use and improved relationship functioning. Yet, community-based treatment programs rarely offer BCT to incoming eligible patients. As reported by providers and administrators in a national survey of treatment programs in the U.S., BCT was viewed as prohibitively labor intensive, due in large measure to its standard conjoint one-couple-at-a-time delivery format. Given the public policy climate that is now emphasizing not only clinical effectiveness, but also economic accountability, an intervention's efficiency (i.e., the ratio of effectiveness to program resources used to provide the service) is a critical factor in decisions by treatment programs to adopt new interventions. Although BCT has well-proven efficacy, the consensus of providers and administrators is that BCT is not efficient.

To address these issues, we have studied couples group formats to deliver BCT. First, in earlier work the PI developed a 10-week BCT group with a number of conjoint sessions added before to prepare couples and afterwards to prevent relapse. While the outcomes were favorable, the added conjoint sessions and the closed group that once begun did not add additional members made it a hard sell for community agencies looking for briefer treatments and typically running ongoing groups with new members added regularly. Second, to overcome these problems, the PI and Co-PI developed a 10-session ongoing BCT group format that has rotating content and rolling admissions in which couples join the group, complete 10 sessions, and "graduate". A major advantage of this ongoing group format for BCT is that it fits with the way other types of groups generally are run in substance abuse programs. It got favorable reviews in provider focus groups and showed promise in a pilot study.

The pilot study with married or cohabiting male drug-abusing patients examined the efficacy of a multi-couple group therapy version of BCT (G-BCT) compared to standard conjoint BCT (S-BCT), and individual-based treatment (group and individual counseling) for the patient only. Results showed G-BCT yielded equivalent outcomes when compared to S-BCT, in terms of reduction in substance use and improved relationship adjustment, but GBCT was less costly to deliver and had superior cost-benefit and cost-effectiveness. Both G-BCT and S-BCT yielded better clinical and cost-outcomes than individual-based treatment. Also, a small-scale evaluation study indicated G-BCT was more likely to be used in community-based treatment programs than S-BCT.

Thus, this proposed study will conduct a randomized clinical trial to examine the clinical effectiveness, in terms of substance use, relationship functioning, and psychosocial adjustment, of Group BCT (G-BCT) versus Standard BCT (S-BCT) for 160 alcoholic patients and their nonsubtance-abusing partners. Given the likely differences in cost of treatment delivery between the 2 interventions, we will also examine the comparative cost-benefit and cost-effectiveness of the 2 intervention packages.

ELIGIBILITY:
Inclusion Criteria:

(a) both members of the couple must be between 18 and 65 years of age; (b) patient must meet Diagnostic and Statistical Manual of Mental Disorders (DSM-IV; American Psychiatric Association, 1994) criteria for current (past 12 months) alcohol dependence and alcohol must be the patient's primary substance of abuse as determined by a clinical algorithm (Fals-Stewart, Stappenbeck et al, 2004); (c) be married to their current partner for at least 1 year or be cohabiting in a stable common-law relationship for 2 years; (d) patient agrees to a goal of abstinence from alcohol and drugs at least for the duration of the 12-week study-based treatment; (e) patient drank in past 60 days; (f) patient agrees to forego other alcoholism counseling except for self-help meetings (e.g., AA) or treatment required for a clinical emergency or clinical deterioration for the duration of the 12-week study-based treatment; (g) no more than 4 months living apart in past year; (h) alcohol dependent patient and partner currently living with each other, i.e., not separated or planning divorce; and (i) both alcohol dependent patient and the relationship partner are willing to participate.

Exclusion Criteria:

a) partner meets DSM-IV criteria for a substance use disorder (other than nicotine) in the last 12 months; (b) patient has dependence on alcohol or other drugs that requires inpatient treatment or medical detoxification (as indicated by daily heavy use or use to prevent or deal with withdrawal symptoms) - after patient has completed detoxification, he or she may be eligible for the study; (c) patient or partner are at immediate risk for suicide or homicide or either made a suicide attempt in past 30 days; and (d) patient or partner meets DSM-IV criteria for a current organic mental disorder, schizophrenia, delusional (paranoid) disorder, or any of the other psychotic disorders. The SCID-IV (SCID; First, Spitzer, Gibbon, & Williams, 1995) will be used to screen out participants with psychosis or thought disorder. Subjects with other disorders, however, will not be excluded. Consistent with general AdCare Hospital services, the AdCare physician can prescribe psychiatric medication (e.g., antidepressants) if necessary. Finally, we also will exclude couples with a recent history (past 3 years) of severe partner violence on a day when drinking or drug use did not occur or if either member of the couple expresses fear that couples therapy may put him or her at risk of violence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Percent days abstinent from alcohol or illicit drugs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J O'Farrell, PhD, Principal Investigator — Harvard Medical School (HMS and HSDM)
Locations (1):
- AdCare Hospital of Worcester, Inc., Worcester, Massachusetts, United States